CLINICAL TRIAL: NCT06920056
Title: A Single Center, Open-label, Fixed Sequence Trial, Investigating the Influence of BGM0504 Injection on Gastric Emptying and Pharmacokinetics of Metformin and Warfarin in Overweight or Obese Participants
Brief Title: A Study of BGM0504 in Overweight or Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGM0504-DDI
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-02

CONDITIONS: Overweight or Obese
MeSH Terms: conditions — Overweight; Obesity | interventions — Acetaminophen; Metformin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paracetamol + Metformin + Warfarin +BGM0504 (Experimental): Participants receive Paracetamol on Day1 and Day70, Metformin on Day4 and Day73, Warfarin on Day7 and Day77.
  Participants receive maintenance dose 10 mg (from D42 to Day 77) with dose escalation starting from 2.5 mg(on Day 14 and Day 21), 5 mg(on Day 28 and Day 35) and then 10 mg BGM0504 administered subcutaneously (SC) once weekly (QW).
  Interventions: Drug: Paracetamol; Drug: Metformin Hydrochloride; Drug: Warfarin; Drug: BGM0504

INTERVENTIONS:
Drug: Paracetamol — oral, postprandial
Drug: Metformin Hydrochloride — Oral , Fasting
Drug: Warfarin — Oral , Fasting
Drug: BGM0504 — Administered SC

SUMMARY:
The purpose of the study is to evaluate the influence of BGM0504 injection on gastric emptying and Pharmacokinetics of metformin and warfarin in overweight or obese participants

ELIGIBILITY:
Inclusion Criteria: √ Have a body mass index (BMI) of greater than or equal to (≥)28 kilogram per square meter (kg/m²) or ≥24 kg/m2 and less than (<) 28 kg/m².

√ Willing and agreeable to commit to the duration of the study and undergo study procedures as instructed by the clinic staff.

Exclusion Criteria: √ History of chronic or acute pancreatitis.

* History of severe drug allergy or specific allergic disease or severe allergies.
* Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2(MEN-2).
* History of malignant tumors [except carcinoma in situ with no recurrence within 5 years (except for malignant melanoma in situ), skin basal cell carcinoma and squamous cell carcinoma].
* Suspected or confirmed history of alcohol or drug abuse;
* Any chronic infections likely to interfere with study conduct or interpretation such as hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) or treponema pallidum (TP).
* Donation or loss of 400 mL or more of blood within 3 months prior to screening, or blood donation during screening or within 3 months after the end of the trial.
* Pregnant or lactating woman.
* Any disorder, unwillingness, or inability not covered by any of the other exclusion criteria, which in the Investigator's opinion, might jeopardize the participant's safety or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC0-t)of Paracetamol | From Day1 to Day72
  Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC0-t) of Paracetamol
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Paracetamol | From Day1 to Day72
  Pharmacokinetics (PK): Maximum observed plasma drug concentration (Cmax) of Paracetamol
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC0-t) of Metformin | From Day4 to Day76
  Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC0-t)of Metformin
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Metformin | From Day4 to Day76
  Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Metformin
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC0-t) of Warfarin | From Day7 to Day84
  Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC0-t) of Warfarin
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Warfarin | From Day7 to Day84
  Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Warfarin

SECONDARY OUTCOMES:
Area Under the Stable-State Concentration Versus Time Curve (AUC0-∞,ss ) of BGM0504 | From Day14 to Day69
  Area Under the Stable-State Concentration Versus Time Curve (AUC0-∞,ss ) of BGM0504
Time to Maximum Concentration (Tmax) of Metformin and Warfarin | From Day1 to Day84
  Time to Maximum Concentration (Tmax) of Metformin and Warfarin
Terminal Half-life (t1/2) of Paracetamol | From Day1 to Day72
  Terminal Half-life (t1/2) of Paracetamol

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Yunnan University of Traditional Chinese Medicine (Yunnan Provincial Hospital of Traditional Chinese Medicine), Kunming, Yunnan, China